CLINICAL TRIAL: NCT05147636
Title: EXtubation With SUctioning or With Positive End-Expiratory Pressure in Intensive Care Unit: a Multicentre Randomised Controlled Trial.
Brief Title: EXtubation With SUctioning or With Positive End-Expiratory Pressure in Intensive Care Unit
Acronym: EXSUPEEP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier de Bourg en Bresse (Other)
Collaborators: Direction Générale de l'Offre de Soins (Other Government); Hospices Civils de Lyon (Other); the EXSUPEEP study was supported by a grant from the French Ministry of Health (MoH-fr) (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: CHB20-001; 2022-A00334-39 (Other: ID RCB/ANSM)
Record Dates: First submitted 2021-11-29; First posted 2021-12-07 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-11

CONDITIONS: Extubation in Intensive Care Unit
Keywords: extubation; intensive care; endotracheal aspiration; positive end expiratory pressure; non invasive ventilation
MeSH Terms: interventions — Airway Extubation; Positive-Pressure Respiration

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PEEP Extubation With Positive End-Expiratory Pressure (Experimental): endo-tracheal aspiration followed by the application of PEEP = 10 cm of H2O, maintained for 3 minutes (reventilation and rest time) and continued until the end of the procedure removal of the extubation
  Interventions: Procedure: Extubation with PEEP
- Aspiration Extubation With SUctioning (Active Comparator): endo-tracheal aspiration concomitant with removal of extubation. Suction is maintained throughout the intubation tube ablation procedure
  Interventions: Procedure: Endotracheal Aspiration

INTERVENTIONS:
Procedure: Extubation with PEEP — No aspiration within the 3 minutes before extubation and extubation with 10cmH2O PEEP
  Arms: PEEP Extubation With Positive End-Expiratory Pressure
Procedure: Endotracheal Aspiration — Aspiration during cuff deflation
  Arms: Aspiration Extubation With SUctioning

SUMMARY:
Extubation in intensive care unit is a risky situation. Its failure is associated with an increase in the duration of mechanical ventilation and high morbidity and mortality.

Our hypothesis is that the extubation procedure associating prior endotracheal aspiration followed by ablation of the intubation probe under the application of a PEEP, would make it possible both to avoid the leakage of secretions towards the lower airways and the alveolar recruitment, compared to extubation with concomitant endotracheal aspiration.

By these mechanisms, this extubation procedure combining prior endotracheal aspiration followed by ablation of the tube under the application of a PEEP, would make it possible to increase the ventilator free days from any mechanical ventilation.

DETAILED DESCRIPTION:
Extubation consists of several distinct phases: obtaining the weaning criteria, succeeding weaning test and then removing the intubation tube.

While the first two stages are the subject of numerous publications, the last one is rarely studied. To reduce the risk of failure of extubation, the scientific societies of intensive care medicine have published recommendations. They relate to patient weaning and weaning testing, but there are no clear recommendations for the procedure for removing the intubation tube.

The ablation of the tube, performed by the chest physiotherapist or nurse, typically involves endotracheal aspiration, from deflation of the cuff to removal of the intubation tube.

The objective is theoretically to prevent the secretions accumulated above the cuff, at the pharyngeal level, from falling into the lower airways.

Laboratory data show that inhalation of secretions appears to be greater during ablation of the tube with concomitant endotracheal aspiration, which creates a reverse pressure gradient, propelling the secretions into the lower airways. The application of Positive Expiratory Pressure during the ablation of the tube would help to combat this phenomenon. At the same time, this Positive Expiratory Pressure could have a beneficial effect on alveolar recruitment.

Recent work proves the non-inferiority of the ablation of the tube with the application of a Positive Expiratory Pressure versus the so-called "reference" method, consisting of endotracheal aspiration during the ablation of the tube.

We wish to conduct a comparative, prospective, randomized, multicenter study comparing extubation with concomitant endotracheal aspiration versus ablation of the intubation tube under the application of a PEEP.

ELIGIBILITY:
Inclusion criteria

Firstly, the decision to extubate must be made by the treating clinicians after having validated that the clinical criteria for weaning are met, namely: according to the international conference consensus on weaning , patients will be considered as ready for an initial SBT as soon as they meet all of the following criteria:

* respiratory rate ≤35 breaths per minute,
* adequate oxygenation defined as pulse oximetry (SpO2 ≥90%) with a fraction of inspired oxygen (FiO2) ≤0.4 or PaO2/FiO2 ≥150 mmHg with positive end-expiratory pressure ≤8 cm H2O,
* hemodynamic stability with no need for vasopressors (or doses ≤0.3 μg/kg/min),
* adequate cough,
* patient awake with a Richmond Agitation-Sedation Scale between +1 and -2

Patients meeting any of the following criteria will be included in the EXSUPEEP trial:

* ICU Hospitalization
* Oro-tracheal intubation
* Mechanical ventilation for more than 24 h
* First extubation procedure during the stay in the including unit
* Consent collected from a relative of the patient. Once it has been verified that the patient meets all the eligibility criteria listed above, the patient may be extubated after a successful SBT and after obtaining consent from the patient or family.

Exclusion criteria

Patients meeting any of the following criteria will be excluded from the EXSUPEEP trial:

* Patients receiving ventilation via tracheostomy.
* Patients with underlying chronic neuromuscular disease
* Patients with severe head injury
* Patients with a decision to withhold and/or withdraw life support
* Patients not affiliated to or beneficiary of any social security scheme.
* Person benefiting from enhanced protection, namely minors, pregnant or nursing women, persons deprived of their liberty by a judicial or administrative decision, persons residing in a healthcare or social establishment, adults under legal protection (safeguard of justice, guardianship or curatorship)
* Inclusion in another research project that interferes with the outcomes of the present study
* Weanability criteria not met within 72 hours following the signing of consent by the relatives.
* Unsuccessful weaning test within 72 hours following the signing of consent by the relatives

Patients with personal NIV or continuous positive airway pressure at home will be included if Pressure Support (PS) and/or PEEP used in the ICU unit are different from the usual settings at home. Regarding infection by SARS-CoV-2 or use of endotracheal tubes with subglottic suction, they do not constitute an exclusion criterion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 425 (Actual)
Dates: Start 2023-03-22 (Actual); Primary Completion 2025-03-19 (Actual); Study Completion 2025-03-19 (Actual)

PRIMARY OUTCOMES:
Ventilator free days at the 28th day | From DZéro to D27
  The primary endpoint is the number of mechanical ventilation-free days (invasive and non-invasive) after the first extubation procedure

SECONDARY OUTCOMES:
Re-intubation rate | 7 days (from Dzéro to D6)
  The re-intubation rate (%) within seven days following the removal of the Extubation Procedure
Cumulated duration of non invasive ventilation (NIV) and High flow oxygenation (HFO) | 7 days (from Dzéro to D6)
  Duration marked in hours , same for NIV and HFO
Proportion of patients with pneumonia and/or atelectasis | within 72 hours ( D2) and within 7 days ( D6)
  radiological assessment of pneumonia and/or atelectasis. A systematic chest radiography is to be done at 72 hours and 7 days after extubation procedure.
Rate of Respiratory acute failure (RAF) | Within 7 days (from Dzéro to D6)
  Percentage of included patients who with clinical RAF after extubation procedure
Lenght of stay in Intensive care unit (ICU) and in hospital | within 28 days
  Marked in days.
Rate of death | Within 28 days (from Dzero to Day 27)
  Whatever the cause of death for included patients

CONTACTS AND LOCATIONS:
Overall Officials: Nicholas SEDILLOT, Principal Investigator — CH Bourg en Bresse
Locations (11):
- France (11):
  - CHU Orléans, Orléans, Orléans
  - CH Annecy Genevois, Annecy
  - CH Victor Dupouy, Argenteuil
  - CH Bourg en Bresse, Bourg-en-Bresse
  - CHU Francois Mitterand, Dijon
  - CHU Michallon, Grenoble
  - HCL Croix Rousse, Lyon
  - HCL Edouard Herriot, Lyon
  - HCL Lyon Sud, Lyon
  - CHU La Miletrie, Poitiers
  - Hopital Nord, Saint-Etienne

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sedillot N, Kallel H, Robine A, Pineda JA, Quenot JP, Servant M, Levrat A, Damieux-Verdeau C, Mezidi M, Thibert N, Bohe J, Ballesteros-Calzado A, Stevic N, Mahi L, Sigaud F, Maisonneuve M, Thiery G, Prat P, Thille AW, Haouat S, Plantefeve G, Decullier E, Rabilloud M, Bernon P, Poncelin Y, Bonnici JC. Applying positive end-expiratory pressure before and during endotracheal tube removal versus extubation with concomitant aspiration: protocol for the randomised controlled multicentre EXSUPEEP trial. BMJ Open. 2025 Feb 13;15(2):e092354. doi: 10.1136/bmjopen-2024-092354. PMID 39947817